CLINICAL TRIAL: NCT04395482
Title: Lung CT Scan Analysis of SARS-CoV2 Induced Lung Injury by Machine Learning: a Multicenter Retrospective Cohort Study.
Brief Title: Lung CT Scan Analysis of SARS-CoV2 Induced Lung Injury
Acronym: TAC-COVID19
Status: Completed | Type: Observational
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Sponsor
Other Study IDs: TAC-COVID19
Record Dates: First submitted 2020-05-18; First posted 2020-05-20 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: covid19
Keywords: Lung injury; sars-covid-2; coronavirus infection
MeSH Terms: conditions — COVID-19; Lung Injury; Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- covid-19 pneumonia related patients: The study aims to collect the highest number possible of lung CT scan images performed in patients with COVID-19, in order to obtain a large sample size that will allow us to characterize the extent of lung injury, the presence of specific patterns of lung alteration, and their potential association with the outcome of patients - in view of assisting the medical staff in better understanding the grade of the severity impairment in these patients which might be potentially candidates to more intensive therapeutic strategies.
  Interventions: Other: Lung CT scan analysis in COVID-19 patients

INTERVENTIONS:
Other: Lung CT scan analysis in COVID-19 patients — This research project will evaluate the morphological characteristics of the lung by CT scan analysis in COVID-19 patients which will be identified as specific patterns using artificial intelligence technology and their impact on outcome.

SUMMARY:
This is a multicenter observational retrospective cohort study that aims to study the morphological characteristics of the lung parenchyma of SARS-CoV2 positive patients identifiable in patterns through artificial intelligence techniques and their impact on patient outcome.

DETAILED DESCRIPTION:
BACKGROUND:

In February, the first case of SARS-CoV2 positive patient was recorded in Lombardy (Italy), a virus capable of causing a severe form of acute respiratory failure called Coronavirus Disease 2019 (COVID-19).

Qualitative assessments of lung morphology have been identified to describe macroscopic characteristics of this infection upon admission and during the hospitalization of patients.

At the moment, there are no studies that have exhaustively described the parenchymal lung damage induced by SARS-CoV2 by quantitative analysis.

The hypothesis of this study is that specific morphological and quantitative alterations of the lung parenchyma assessed by means of CT scan in patients suffering from severe respiratory insufficiency induced by SARS-CoV2 may have an impact on the severity of the degree of alteration of the respiratory exchanges (oxygenation and clearance of the CO2) and have an impact on patient outcome.

The presence of characteristic lung morphological patterns assessed by CT scan could allow the recognition of specific patient clusters who can benefit from intensive treatment differently, making a significant contribution to stratifying the severity of patients and their risk of mortality.

This is an exploratory clinical descriptive study of lung CT images in a completely new patient population who are nucleic acid amplification test confirmed SARS-CoV2 positive.

SAMPLE SIZE (n. patients):

The study will collect all patients with the inclusion criteria; a total of 500 patients are expected to be collected.

About 80 patients will be enrolled for each local experimental center.

The following patient data will be analyzed:

* blood gas analytical data assigned to the CT scan, checks performed upon entering the hospital, at the time of performing the CT scan, admission to intensive care and 7 days after entry
* patient characteristics such as age, gender and body mass index (BMI)
* comorbidity
* presence of organ dysfunction with the Sequential Organ Failure Assessment (SOFA)
* laboratory data relating to hospital admission and symptoms prior to hospitalization.
* ventilator and hemodynamic parameters upon entering the hospital, at the time of carrying out the CT scan, upon admission to intensive care and 7 days after entry.

The machine learning approach of lung CT scan analysis will aim at evaluating:

1. Quantitative and qualitative lung alterations;
2. The stratification of such morphological characteristics in specific morphological lung clusters identified by the means of artificial intelligence using deep learning algorithms.

ETHICAL ASPECTS:

The lung CT scan images will be collected and anonymized. Images will be subsequently sent by University of Milano-Bicocca Institutional google drive account to the University of Pennsylvania, Department of Anesthesiology and Critical Care and the Department of Radiology in a deidentified format for advanced quantitative analysis taking advantage of artificial intelligence using deep learning algorithms.

The data will be collected in a pseudo-anonymous way through paper Case Report Form (CRF) and analyzed by the scientific coordinator of the project.

Given the retrospective nature of the study and in the presence of technical difficult in obtaining an informed consent of patients in this period of pandemic emergency, informed consent will be waived.

STATISTICAL ANALYSIS:

Continuous data will be expressed as mean ± standard deviation or median and interquartile range, according to data distribution that will be evaluated by the Shapiro-Wilk test. Categorical variables will be expressed as proportions (frequency).

The deep learning segmentation algorithm will segment the lung parenchyma from the entire CT lung. Lung volume, lung weight and opacity intensity distribution analysis will be applied. Second, clustering analysis to stratify the patients will be performed. Both an intensity and a spatial clustering algorithm will be tested. Third, a model will be trained to predict the injury progression using the images and all other patient data. Statistical significance will be considered in the presence of a p<0.05 (two-tailed).

ELIGIBILITY:
Inclusion Criteria (COVID-19 cohort):

* Patients 18 years old or above;
* Positive confirmation with nucleic acid amplification test or serology of SARS-CoV2 by naso-pharyngeal swab, bronchoaspirate sample or bronchoalveolar lavage;
* Lung CT scan performed within 7 days of hospital admission;

Inclusion criteria (ARDS cohort):

* Patients above 18 years old or above;
* Patients admitted to the hospital with a diagnosis of ARDS according to the Berlin criteria;
* Lung CT scan performed within 7 days of ARDS diagnosis;

Exclusion criteria (ARDS cohort):

● Positive confirmation with nucleic acid amplification test or serology of SARS-CoV2 by naso-pharyngeal swab, bronchoaspirate sample or bronchoalveolar lavage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The goal is to collect as many lung CT scan images as possible in patients with COVID-19; according to the preliminary evaluation estimate, a total of 500 patients are expected to be collected.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2020-05-07 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
A qualitative analysis of parenchymal lung damage induced by COVID-19 | Until patient discharge from the hospital (approximately 6 months)
  Describe the parenchymal lung damage induced by COVID-19 through a qualitative analysis with chest CT through artificial intelligence techniques.
A quantitative analysis of parenchymal lung damage induced by COVID-19 | Until patient discharge from the hospital (approximately 6 months)
  Describe the parenchymal lung damage induced by COVID-19 through a quantitative analysis with chest CT through artificial intelligence techniques.

SECONDARY OUTCOMES:
The potential impact of parenchymal morphological CT scans in patients with severe moderate respiratory failure. | Until patient discharge from the hospital (approximately 6 months)
  The potential impact of parenchymal morphological CT scans in patients with severe moderate respiratory failure assessed as intensive care mortality.
The potential impact of parenchymal morphological CT scans in patients with severe moderate respiratory failure. | Until patient discharge from the hospital (approximately 6 months)
  The potential impact of parenchymal morphological CT scans in patients with severe moderate respiratory failure assessed as hospital mortality.
The potential impact of parenchymal morphological CT scans in patients with severe moderate respiratory failure. | Until patient discharge from the hospital (approximately 6 months)
  The potential impact of parenchymal morphological CT scans in patients with severe moderate respiratory failure assessed as days free from mechanical ventilation.
Automated segmentation of lung scans of patients with COVID-19 and ARDS. | Until patient discharge from the hospital (approximately 6 months)
  The hypothesis is that the uso of deep neural network models for lung segmentation in Acute Respiratory Distress Syndrome (ARDS) in animal models and Chronic Obstructive Pulmonary Disease (COPD) in patients that could be applied to self-segment the lungs of COVID-19 patients through a learning transfer mechanism with artificial intelligence.
Knowledge of chest CT features in COVID-19 patients and their detail through the use of machine learning and other quantitative techniques. | Until patient discharge from the hospital (approximately 6 months)
  Expand the knowledge of chest CT features in COVID-19 patients and their detail through the use of machine learning and other quantitative techniques comparing CT patterns of COVID-19 patients to those of patients with ARDS.
The ability within which the analysis of artificial intelligence that uses deep learning models can be used to predict clinical outcomes | Until patient discharge from the hospital (approximately 6 months)
  Determine the capacity within which the artificial intelligence analysis that uses deep learning models can be used to predict clinical outcomes from the analysis of the characteristics of the chest CT obtained within 7 days of hospital admission; combining quantitative CT data with clinical data.

CONTACTS AND LOCATIONS:
Locations (8):
- Italy (7):
  - Ospedale Papa Giovanni XXIII, Bergamo
  - Policlinico San Marco-San Donato group, Bergamo
  - Azienda Ospedaliero-Universitaria di Ferrara, Ferrara
  - ASST di Lecco Ospedale Alessandro Manzoni, Lecco
  - ASST Melegnano-Martesana, Ospedale Santa Maria delle Stelle, Melzo
  - ASST Monza, Monza
  - AUSL Romagna-Ospedale Infermi di Rimini, Rimini
- Istituto per la Sicurezza Sociale-Ospedale della Repubblica di San Marino, San Marino, San Marino

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grasselli G, Pesenti A, Cecconi M. Critical Care Utilization for the COVID-19 Outbreak in Lombardy, Italy: Early Experience and Forecast During an Emergency Response. JAMA. 2020 Apr 28;323(16):1545-1546. doi: 10.1001/jama.2020.4031. No abstract available. PMID 32167538
- [Background] Remuzzi A, Remuzzi G. COVID-19 and Italy: what next? Lancet. 2020 Apr 11;395(10231):1225-1228. doi: 10.1016/S0140-6736(20)30627-9. Epub 2020 Mar 13. PMID 32178769
- [Background] Dong E, Du H, Gardner L. An interactive web-based dashboard to track COVID-19 in real time. Lancet Infect Dis. 2020 May;20(5):533-534. doi: 10.1016/S1473-3099(20)30120-1. Epub 2020 Feb 19. No abstract available. PMID 32087114
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Background] Zhou S, Wang Y, Zhu T, Xia L. CT Features of Coronavirus Disease 2019 (COVID-19) Pneumonia in 62 Patients in Wuhan, China. AJR Am J Roentgenol. 2020 Jun;214(6):1287-1294. doi: 10.2214/AJR.20.22975. Epub 2020 Mar 5. PMID 32134681
- [Background] Xiong Y, Sun D, Liu Y, Fan Y, Zhao L, Li X, Zhu W. Clinical and High-Resolution CT Features of the COVID-19 Infection: Comparison of the Initial and Follow-up Changes. Invest Radiol. 2020 Jun;55(6):332-339. doi: 10.1097/RLI.0000000000000674. PMID 32134800
- [Background] Salehi S, Abedi A, Balakrishnan S, Gholamrezanezhad A. Coronavirus Disease 2019 (COVID-19): A Systematic Review of Imaging Findings in 919 Patients. AJR Am J Roentgenol. 2020 Jul;215(1):87-93. doi: 10.2214/AJR.20.23034. Epub 2020 Mar 14. PMID 32174129
- [Background] Dai WC, Zhang HW, Yu J, Xu HJ, Chen H, Luo SP, Zhang H, Liang LH, Wu XL, Lei Y, Lin F. CT Imaging and Differential Diagnosis of COVID-19. Can Assoc Radiol J. 2020 May;71(2):195-200. doi: 10.1177/0846537120913033. Epub 2020 Mar 4. PMID 32129670
- [Background] Li Y, Xia L. Coronavirus Disease 2019 (COVID-19): Role of Chest CT in Diagnosis and Management. AJR Am J Roentgenol. 2020 Jun;214(6):1280-1286. doi: 10.2214/AJR.20.22954. Epub 2020 Mar 4. PMID 32130038
- [Background] Xie X, Zhong Z, Zhao W, Zheng C, Wang F, Liu J. Chest CT for Typical Coronavirus Disease 2019 (COVID-19) Pneumonia: Relationship to Negative RT-PCR Testing. Radiology. 2020 Aug;296(2):E41-E45. doi: 10.1148/radiol.2020200343. Epub 2020 Feb 12. PMID 32049601
- [Background] Ai T, Yang Z, Hou H, Zhan C, Chen C, Lv W, Tao Q, Sun Z, Xia L. Correlation of Chest CT and RT-PCR Testing for Coronavirus Disease 2019 (COVID-19) in China: A Report of 1014 Cases. Radiology. 2020 Aug;296(2):E32-E40. doi: 10.1148/radiol.2020200642. Epub 2020 Feb 26. PMID 32101510
- [Background] Fang Y, Zhang H, Xie J, Lin M, Ying L, Pang P, Ji W. Sensitivity of Chest CT for COVID-19: Comparison to RT-PCR. Radiology. 2020 Aug;296(2):E115-E117. doi: 10.1148/radiol.2020200432. Epub 2020 Feb 19. No abstract available. PMID 32073353
- [Background] Bai HX, Hsieh B, Xiong Z, Halsey K, Choi JW, Tran TML, Pan I, Shi LB, Wang DC, Mei J, Jiang XL, Zeng QH, Egglin TK, Hu PF, Agarwal S, Xie FF, Li S, Healey T, Atalay MK, Liao WH. Performance of Radiologists in Differentiating COVID-19 from Non-COVID-19 Viral Pneumonia at Chest CT. Radiology. 2020 Aug;296(2):E46-E54. doi: 10.1148/radiol.2020200823. Epub 2020 Mar 10. PMID 32155105
- [Background] Pan F, Ye T, Sun P, Gui S, Liang B, Li L, Zheng D, Wang J, Hesketh RL, Yang L, Zheng C. Time Course of Lung Changes at Chest CT during Recovery from Coronavirus Disease 2019 (COVID-19). Radiology. 2020 Jun;295(3):715-721. doi: 10.1148/radiol.2020200370. Epub 2020 Feb 13. PMID 32053470
- [Background] Chung M, Bernheim A, Mei X, Zhang N, Huang M, Zeng X, Cui J, Xu W, Yang Y, Fayad ZA, Jacobi A, Li K, Li S, Shan H. CT Imaging Features of 2019 Novel Coronavirus (2019-nCoV). Radiology. 2020 Apr;295(1):202-207. doi: 10.1148/radiol.2020200230. Epub 2020 Feb 4. PMID 32017661
- [Background] Bernheim A, Mei X, Huang M, Yang Y, Fayad ZA, Zhang N, Diao K, Lin B, Zhu X, Li K, Li S, Shan H, Jacobi A, Chung M. Chest CT Findings in Coronavirus Disease-19 (COVID-19): Relationship to Duration of Infection. Radiology. 2020 Jun;295(3):200463. doi: 10.1148/radiol.2020200463. Epub 2020 Feb 20. PMID 32077789
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Shi H, Han X, Jiang N, Cao Y, Alwalid O, Gu J, Fan Y, Zheng C. Radiological findings from 81 patients with COVID-19 pneumonia in Wuhan, China: a descriptive study. Lancet Infect Dis. 2020 Apr;20(4):425-434. doi: 10.1016/S1473-3099(20)30086-4. Epub 2020 Feb 24. PMID 32105637
- [Background] Guo L, Wei D, Zhang X, Wu Y, Li Q, Zhou M, Qu J. Clinical Features Predicting Mortality Risk in Patients With Viral Pneumonia: The MuLBSTA Score. Front Microbiol. 2019 Dec 3;10:2752. doi: 10.3389/fmicb.2019.02752. eCollection 2019. PMID 31849894
- [Background] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Background] Chen N, Zhou M, Dong X, Qu J, Gong F, Han Y, Qiu Y, Wang J, Liu Y, Wei Y, Xia J, Yu T, Zhang X, Zhang L. Epidemiological and clinical characteristics of 99 cases of 2019 novel coronavirus pneumonia in Wuhan, China: a descriptive study. Lancet. 2020 Feb 15;395(10223):507-513. doi: 10.1016/S0140-6736(20)30211-7. Epub 2020 Jan 30. PMID 32007143
- [Background] Yang X, Yu Y, Xu J, Shu H, Xia J, Liu H, Wu Y, Zhang L, Yu Z, Fang M, Yu T, Wang Y, Pan S, Zou X, Yuan S, Shang Y. Clinical course and outcomes of critically ill patients with SARS-CoV-2 pneumonia in Wuhan, China: a single-centered, retrospective, observational study. Lancet Respir Med. 2020 May;8(5):475-481. doi: 10.1016/S2213-2600(20)30079-5. Epub 2020 Feb 24. PMID 32105632
- [Background] Ki M; Task Force for 2019-nCoV. Epidemiologic characteristics of early cases with 2019 novel coronavirus (2019-nCoV) disease in Korea. Epidemiol Health. 2020;42:e2020007. doi: 10.4178/epih.e2020007. Epub 2020 Feb 9. PMID 32035431
- [Derived] Rezoagli E, Xin Y, Signori D, Sun W, Gerard S, Delucchi KL, Magliocca A, Vitale G, Giacomini M, Mussoni L, Montomoli J, Subert M, Ponti A, Spadaro S, Poli G, Casola F, Herrmann J, Foti G, Calfee CS, Laffey J, Bellani G, Cereda M; CT-COVID19 Multicenter Study Group. Phenotyping COVID-19 respiratory failure in spontaneously breathing patients with AI on lung CT-scan. Crit Care. 2024 Aug 5;28(1):263. doi: 10.1186/s13054-024-05046-3. PMID 39103945
- See also: Related Info — http://coronavirus.jhu.edu/map.html
- See also: Related Info — http://www.cnr.it/it/nota-stampa/n-9281/analisi-numerica-dei-dati-relativi-alla-diffusione-del-covid-19-in-italia-e-nel-mondo